CLINICAL TRIAL: NCT00461656
Title: Prospective, Randomized, Double-blind Comparison of 5 % Against 1.25 % Povidone-iodine Solution as Preoperative Antisepsis for Strabismus Surgery in Young Children
Brief Title: Povidone-iodine Antisepsis for Strabismus Surgery
Acronym: PASS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); University Medicine Greifswald (Other); Free University Medical Center (Other); Leiden University Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Rotterdam Eye Hospital (Unknown); Laurentius Hospital Roermond (Unknown); Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Prof. H.J. Simonsz M.D., Erasmus Medical Center Rotterdam
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ABR 14357
Record Dates: First submitted 2007-04-17; First posted 2007-04-18 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2011-07

CONDITIONS: Strabismus; Surgery; Endophthalmitis
Keywords: Antiseptic; Povidone-Iodine
MeSH Terms: conditions — Strabismus; Endophthalmitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Preoperative conjunctival irrigation with 5% or 1.25% PI — Before initiation of surgery, children will have their conjunctival fornices irrigated with 5 ml PI 5% or with 5 ml PI 1.25%

SUMMARY:
The purpose of this study is to compare the efficacy of 5 % vs. 1.25 % povidone-iodine (PI) as preoperative antiseptic prior to strabismus surgery in children as a prophylaxis of endophthalmitis. Given the low rate of endophthalmitis the conjunctival bacterial flora rate is used as surrogate marker to determine the effectiveness of topical PI in reducing or eliminating bacteria from the ocular surface at the time of the surgery. Secondary objective is a reduction of the incidence of postoperative endophthalmitis after strabismus surgery in young children.

DETAILED DESCRIPTION:
Background: Endophthalmitis after strabismus surgery in young children leads to blindness and loss of the affected eye. It is caused by conjunctival bacteria. PI solutions between 1% and 5% reduce the number of bacteria on the conjunctiva. The concentration used varies widely among clinics, from 1% to 5%. In vitro studies have shown that PI is paradoxically more effective at lower concentration, but in cataract surgery in elderly, 1% PI has been shown to be less effective than 5% PI. Dilution by tear fluid or binding of PI to proteins in tear fluid may lower its effectiveness. Since endophthalmitis after strabismus surgery especially affects young children and the bacterial flora of the conjunctiva in children is different from that in adults, the cataract PI study should be repeated in young children operated for strabismus.

Objective: To compare the efficacy of 5 % vs. 1.25 % povidone-iodine (PI) as preoperative antiseptic prior to strabismus surgery in children as a prophylaxis of endophthalmitis. Given the low rate of endophthalmitis the conjunctival bacterial flora rate is used as surrogate marker to determine the effectiveness of topical PI in reducing or eliminating bacteria from the ocular surface at the time of the surgery.

Design: The study is a multi-centre, prospective, randomized-controlled, parallel-groups, assessor-blind (microbiological assessments), investigator-initiated trial.

Study population: All children under 6 years of age attending the 15 participating clinics for routine strabismus surgery will be eligible for the study at the point that a strabismus operation is planned. The clinics (5 Dutch, 10 German) will each recruit approximately 20 patients. The minimum sample size is 2 x 100 patients.

Intervention: Diluted PI, 1.25% or 5%, will be prepared in a sterile fashion, and distributed in single-use dispensers. These will be coded for randomization. Before initiation of surgery, children randomized to the 5% PI group will have their conjunctival fornices irrigated with 5 ml PI 5%. Children randomized to the 1.25% PI group will have their conjunctival fornices irrigated with 5 ml PI 1.25%. Conjunctiva cultures for aerobic and anaerobic bacteria will be obtained (1) after general anesthesia has been established, (2) 5-10 min after PI irrigation, (3) after reattachment of the eye muscles and (4) after closing the conjunctiva with sutures.

Primary outcome: The difference in the mean numbers of bacterial colony forming units (CFUs) from pre-irrigation (l) to post-irrigation with PI (2-4).

Secondary outcome: Iodine excretion after surgery, assessed as urine iodine concentration per creatinine clearance.

Postoperative erosion of the cornea and corneal oedema. Both of these have been described as side-effects of PI use.

Nature and extent of the burden and risks associated with participation:

Risks are limited to the act of taking the four bacterial cultures, as both 1.25% PI and 5% PI are approved preoperative antiseptic applications of PI and both are used, rather indiscriminately, by the university departments of ophthalmology participating in the study.

ELIGIBILITY:
Inclusion Criteria:

Children attending for routine strabismus surgery are eligible for the study. Criteria for inclusion:

1. Children < 6 years of age
2. undergoing surgery for strabismus for the first time, including any recession and/or resection surgery of the medial and/or lateral rectus muscles.
3. willing to take part in all aspects of the study with written informed consent on the study participation of the child provided by the parents.

Exclusion Criteria:

1. Any history or current condition of hypersensitivity to iodine
2. Children on topical antibiotic within the last 30 days
3. Children with signs of acute conjunctivitis, blepharitis, dacryocystitis or respiratory infection within the last 30 days
4. Children with asthma or similar chronic, obstructive pulmonary disorder
5. Insufficiently treated amblyopia, i.e. a difference between the visual acuities of both eyes larger than 1 LogMARline.
6. Neurological or psychiatric disorder, medication, other eye disorder, decreased visual acuity caused by brain damage or trauma.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The difference in the mean numbers of bacterial colony forming units from pre-irrigation to post-irrigation with PI. | Cultures taken during surgery, evaluated within 2 days postoperatively

SECONDARY OUTCOMES:
Iodine excretion after surgery, assessed as urine iodine concentration per creatinine clearance. | 24 hours postoperatively
Postoperative erosion of the cornea and corneal oedema. | within 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Huibert J Simonsz, MD PhD, Principal Investigator — Erasmus Medical Center; Herminia Miño de Kaspar, PhD, Principal Investigator — Universitäts-Augenklinik Ludwig-Maximilian University Munich Germany
Locations (9):
- Germany (3):
  - Ernst Moritz Arndt University, Greifswald
  - Universitäts-Augenklinik, Magdeburg
  - Universitäts-Augenklinik Ludwig-Maximilian University, Munich
- Netherlands (6):
  - Dept. Ophthalmology Free University Medical Center, Amsterdam
  - Dept. Ophthalmology Academical Medical Center, Amsterdam
  - Dept. Ophthalmology, Leiden
  - Dept. of Ophthalmology St. Laurentius Ziekenhuis, Roermond
  - Rotterdam Eye Hospital, Rotterdam
  - Dept. of Ophthalmology Erasmus Medical Center, Rotterdam

REFERENCES:
- [Background] Anderson RL, Vess RW, Carr JH, Bond WW, Panlilio AL, Favero MS. Investigations of intrinsic Pseudomonas cepacia contamination in commercially manufactured povidone-iodine. Infect Control Hosp Epidemiol. 1991 May;12(5):297-302. doi: 10.1086/646342. PMID 1865100
- [Background] Apt L, Isenberg S, Yoshimori R, Paez JH. Chemical preparation of the eye in ophthalmic surgery. III. Effect of povidone-iodine on the conjunctiva. Arch Ophthalmol. 1984 May;102(5):728-9. doi: 10.1001/archopht.1984.01040030584025. PMID 6721765
- [Background] Bannerman TL, Rhoden DL, McAllister SK, Miller JM, Wilson LA. The source of coagulase-negative staphylococci in the Endophthalmitis Vitrectomy Study. A comparison of eyelid and intraocular isolates using pulsed-field gel electrophoresis. Arch Ophthalmol. 1997 Mar;115(3):357-61. doi: 10.1001/archopht.1997.01100150359008. PMID 9076208
- [Background] Berkelman RL, Holland BW, Anderson RL. Increased bactericidal activity of dilute preparations of povidone-iodine solutions. J Clin Microbiol. 1982 Apr;15(4):635-9. doi: 10.1128/jcm.15.4.635-639.1982. PMID 7040461
- [Background] Binder CA, Mino de Kaspar H, Klauss V, Kampik A. [Preoperative infection prophylaxis with 1% polyvidon-iodine solution based on the example of conjunctival staphylococci]. Ophthalmologe. 1999 Oct;96(10):663-7. doi: 10.1007/s003470050471. German. PMID 10552160
- [Background] Caldwell DR, Kastl PR, Cook J, Simon J. Povidone-iodine: its efficacy as a preoperative conjunctival and periocular preparation. Ann Ophthalmol. 1984 Jun;16(6):577, 580. PMID 6611102
- [Background] Carothers TS, Coats DK, McCreery KM, Rossman SN, Wilson P, Wu TG, Paysse EA. Quantification of incidental needle and suture contamination during strabismus surgery. Binocul Vis Strabismus Q. 2003;18(2):75-9. PMID 12765540
- [Background] Ciulla TA, Starr MB, Masket S. Bacterial endophthalmitis prophylaxis for cataract surgery: an evidence-based update. Ophthalmology. 2002 Jan;109(1):13-24. doi: 10.1016/s0161-6420(01)00899-5. PMID 11772573
- [Background] Davis GH, Finlayson N, Kemp R. Dilution of povidone-iodine. Med J Aust. 1985 Sep 30;143(7):321. doi: 10.5694/j.1326-5377.1985.tb123038.x. No abstract available. PMID 4046931
- [Background] Dereklis DL, Bufidis TA, Tsiakiri EP, Palassopoulos SI. Preoperative ocular disinfection by the use of povidone-iodine 5%. Acta Ophthalmol (Copenh). 1994 Oct;72(5):627-30. doi: 10.1111/j.1755-3768.1994.tb07191.x. PMID 7887164
- [Background] Ferguson AW, Scott JA, McGavigan J, Elton RA, McLean J, Schmidt U, Kelkar R, Dhillon B. Comparison of 5% povidone-iodine solution against 1% povidone-iodine solution in preoperative cataract surgery antisepsis: a prospective randomised double blind study. Br J Ophthalmol. 2003 Feb;87(2):163-7. doi: 10.1136/bjo.87.2.163. PMID 12543744
- [Background] Grimes SR, Hollsten D, Nauschuetz WF, Whiddon RG, Trevino SB. Effect of povidone-iodine irrigation on the preoperative chemical preparation of the eye. Mil Med. 1992 Mar;157(3):111-3. PMID 1603399
- [Background] Katosova LK. [The features of Haemophilus influenza and Streptococcus pneumoniae carriage and the comparative characteristics of strains isolated from healthy children and from patients with acute and chronic respiratory infections]. Zh Mikrobiol Epidemiol Immunobiol. 1994 Aug-Sep;Suppl 1:55-60. Russian. PMID 7856352
- [Background] Khashu M, Chessex P, Chanoine JP. Iodine overload and severe hypothyroidism in a premature neonate. J Pediatr Surg. 2005 Feb;40(2):E1-4. doi: 10.1016/j.jpedsurg.2004.10.028. PMID 15750908
- [Background] Lacey RW, Catto A. Action of povidone-iodine against methicillin-sensitive and -resistant cultures of Staphylococcus aureus. Postgrad Med J. 1993;69 Suppl 3(818):S78-83. PMID 8290463
- [Background] Mino de Kaspar H, Chang RT, Singh K, Egbert PR, Blumenkranz MS, Ta CN. Prospective randomized comparison of 2 different methods of 5% povidone-iodine applications for anterior segment intraocular surgery. Arch Ophthalmol. 2005 Feb;123(2):161-5. doi: 10.1001/archopht.123.2.161. PMID 15710810
- [Background] Olitsky SE, Vilardo M, Awner S, Reynolds JD. Needle sterility during strabismus surgery. J AAPOS. 1998 Jun;2(3):151-2. doi: 10.1016/s1091-8531(98)90006-4. PMID 10532751
- [Background] Prince HN, Nonemaker WS, Norgard RC, Prince DL. Drug resistance studies with topical antiseptics. J Pharm Sci. 1978 Nov;67(11):1629-31. doi: 10.1002/jps.2600671134. PMID 712607
- [Background] Recchia FM, Baumal CR, Sivalingam A, Kleiner R, Duker JS, Vrabec TR. Endophthalmitis after pediatric strabismus surgery. Arch Ophthalmol. 2000 Jul;118(7):939-44. PMID 10900107
- [Background] Roberts SM, Severin GA, Lavach JD. Antibacterial activity of dilute povidone-iodine solutions used for ocular surface disinfection in dogs. Am J Vet Res. 1986 Jun;47(6):1207-10. PMID 3729119
- [Background] Singer TR, Isenberg SJ, Apt L. Conjunctival anaerobic and aerobic bacterial flora in paediatric versus adult subjects. Br J Ophthalmol. 1988 Jun;72(6):448-51. doi: 10.1136/bjo.72.6.448. PMID 3390421
- [Background] Speaker MG, Milch FA, Shah MK, Eisner W, Kreiswirth BN. Role of external bacterial flora in the pathogenesis of acute postoperative endophthalmitis. Ophthalmology. 1991 May;98(5):639-49; discussion 650. doi: 10.1016/s0161-6420(91)32239-5. PMID 2062496
- [Background] Speaker MG, Menikoff JA. Prophylaxis of endophthalmitis with topical povidone-iodine. Ophthalmology. 1991 Dec;98(12):1769-75. doi: 10.1016/s0161-6420(91)32052-9. PMID 1775308
- [Background] Zamora JL. Chemical and microbiologic characteristics and toxicity of povidone-iodine solutions. Am J Surg. 1986 Mar;151(3):400-6. doi: 10.1016/0002-9610(86)90477-0. PMID 3513654
- [Background] Zamora JL, Price MF, Chuang P, Gentry LO. Inhibition of povidone-iodine's bactericidal activity by common organic substances: an experimental study. Surgery. 1985 Jul;98(1):25-9. PMID 4012604